CLINICAL TRIAL: NCT04315025
Title: Safety Issues of Peribulbar Injection of Umbilical Cord Mesenchymal Stem Cell (UC-MSC) in Patients With Retinitis Pigmentosa
Brief Title: Safety Issues of Peribulbar Injection of UC-MSC in Patients With Retinitis Pigmentosa
Acronym: RP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT/RP/02/2018
Record Dates: First submitted 2020-03-08; First posted 2020-03-19 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-03

CONDITIONS: Retinitis Pigmentosa
Keywords: Allogeneic Mesenchymal Stem Cell; Umbilical Cord Mesenchymal Stem Cell; Conditioned Medium; Allogeneic Umbilical Cord Mesenchymal Stem Cell
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Culture Media, Conditioned

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conditioned Medium (CM) (Active Comparator): a total 2 ml volume of Conditioned Medium derived Umbilical Cord Mesenchymal Stem Cell will be injected by peribulbar
  Interventions: Biological: Conditioned Medium (CM)
- UC-MSC + NaCl (Active Comparator): 1.8 ml cell preparations are suspended in physiological NaCl until it reaches a total of 2 ml volume of cell suspension. Umbilical Cord Mesenchymal Stem Cell (UC-MSC) suspension will be injected by peribulbar
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cell (UC-MSC)
- UC-MSC+CM (Active Comparator): 1.8 ml cell preparations are suspended in Conditioned Medium (CM) until it reaches total of 2 ml volume of cell suspension. Umbilical Cord Mesenchymal Stem Cell (UC-MSC) + Conditioned Medium (CM) suspension will be injected by peribulbar
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cell (UC-MSC); Biological: Conditioned Medium (CM)

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cell (UC-MSC) — Umbilical Cord Mesenchymal Stem Cell (UC-MSC) injected by peribulbar
  Arms: UC-MSC + NaCl; UC-MSC+CM
Biological: Conditioned Medium (CM) — Conditioned Medium (CM) injected by peribulbar
  Arms: Conditioned Medium (CM); UC-MSC+CM

SUMMARY:
The study will perform UC-MSCs and CM transplantation. The first group will be injected by UCMSC+NaCl. the 2nd group will be injected by UC-MSC+CM. the 3rd group will be injected by CM. Each group consists of 6 subjects. all groups will be transplanted via peribulbar route. the dosage of UC-MSC is 1 million cells for each subject. All groups will be observed until 6 months.

DETAILED DESCRIPTION:
The eyes which will give the transplant should be given an aseptic and antiseptic technique to prevent the contamination from the inside and outside. Sterile cover attached to other parts of the face except for the eyes. 1.8 ml cell preparations are suspended in physiological NaCl until it reaches a total of 2 ml volume of cell suspension (for UC-MSC + NaCl group). Stem cell suspension will be injected by peribulbar and if the injection was done, patients will be given a quinolone antibiotic. On day 1st and day 7th after therapy, patients will be observed the presence of infection, inflammation, and increasing of eye pressure. On day 7th, day 30th, and day 90th after therapy, patients will do a visual field test, visual acuity test, electroretinography, funduscopy, and Optical Coherence Tomography examination. The observation results will be written in the observation table and analyzed by a statistic. After the data was completed, then make a discussion, conclusion, and suggestion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Visual field defects at initial examination with Humhprey perimetry are between 25% to 50%
* Willing to sign informed consent as research subjects
* Willing to do peribulbar injection with mesenchymal stem cells isolated from umbilical cord tissue
* Willing to do visual field checks with Humphrey's perimetry, vision tests with Snellen boards, Optical Coherrent Tomography (OCT) examinations, electroretinogram examinations and fill out a quality of life questionnaire

Exclusion Criteria:

* Pregnant or nursing women
* Positive result of HIV test
* Have a history of eye tumors
* In immunosuppressive treatment or other drugs that can affect the growth of transplanted stem cells
* Have another eye disease such as diabetic retinopathy, uveitis, cataract, and glaucoma
* Do not come to control according to the schedule determined by the researcher (loss to follow up)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-07 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Visual Acuity Test | 1 week after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Acuity Test | 1 month after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Acuity Test | 3 months after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Field Test | 1 week after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humprey's perimetry.
Visual Field Test | 1 month after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humprey's perimetry.
Visual Field Test | 3 months after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humprey's perimetry.
Funduscopy | 1 week after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Funduscopy | 1 month after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Funduscopy | 3 months after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Electrorectinography | 1 week after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Electrorectinography | 1 month after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Electrorectinography | 3 months after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Optical Coherence Tomography (OCT) | 1 week after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities
Optical Coherence Tomography (OCT) | 1 month after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities
Optical Coherence Tomography (OCT) | 3 months after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities
Angiography | 1 week after injection
  a process of taking photos of the retina by injecting fluorescent to get a bleeding location on the retina.
Angiography | 1 month after injection
  a process of taking photos of the retina by injecting fluorescent to get a bleeding location on the retina.
Angiography | 3 months after injection
  a process of taking photos of the retina by injecting fluorescent to get a bleeding location on the retina.

CONTACTS AND LOCATIONS:
Overall Officials: dr Cosmos O Mangunsong, Sp.M, Principal Investigator — Gadjah Mada University, Faculty of Medicine; Professor dr. Yohanes W Wirohadidjojo, Sp.KK(K), PhD, Study Director — Gadjah Mada University, Faculty of Medicine; Bayu W Putera, S.Si, M.Kes, Study Director — Prodia Stem Cell Indonesia; dr Bayu M Sasongko, Sp.M, PhD, Study Director — Gadjah Mada University, Faculty of Medicine; dr Melita S Djaja, Sp.M, Study Chair — Jakarta Eye Center; dr Amyra D Costa, Study Chair — Jakarta Eye Center; Rima Haifa, B.Sc, Study Chair — Prodia StemCell Indonesia
Locations (2):
- Indonesia (2):
  - Jakarta Eye Center Hospital, Jakarta, DKI Jakarta
  - Sardjito Hospital, Yogyakarta, Special Region